CLINICAL TRIAL: NCT03570749
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Operationally Seamless, Adaptive Phase 2/3 Study to Evaluate the Efficacy and Safety of Baricitinib in Adult Patients With Severe or Very Severe Alopecia Areata
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Severe or Very Severe Alopecia Areata
Acronym: BRAVE-AA1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16582; I4V-MC-JAHO (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 4 Milligram (mg) Baricitinib Phase 2 (Experimental): Participants received one 4 mg Baricitinib tablet administered orally, every day (QD) and two placebo tablets (QD) administered orally to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib Phase 2 (Experimental): Participants received one 2 mg Baricitinib tablet administered orally QD, and two placebo tablets administered orally QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 1 mg Baricitinib Phase 2 (Experimental): Participants received one 1 mg Baricitinib tablet administered orally QD, and two placebo tablets administered orally QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo Phase 2 (Placebo Comparator): Participants received three placebo tablets administered orally QD to maintain the blind.
  Interventions: Drug: Placebo
- 4 mg Baricitinib Phase 3 (Experimental): Participants received one 4 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2 mg Baricitinib Phase 3 (Experimental): Participants received one 2 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain the blind.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo Phase 3 (Placebo Comparator): Participants received two placebo tablets administered orally QD.
  Interventions: Drug: Placebo
- Open-Label Addenda Baricitinib High Dose (Experimental): Baricitinib will be administered orally during the open-label addenda.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 1 mg Baricitinib Phase 2; 2 mg Baricitinib Phase 2; 2 mg Baricitinib Phase 3; 4 Milligram (mg) Baricitinib Phase 2; 4 mg Baricitinib Phase 3; Open-Label Addenda Baricitinib High Dose
Drug: Placebo — Administered orally.
  Arms: 1 mg Baricitinib Phase 2; 2 mg Baricitinib Phase 2; 2 mg Baricitinib Phase 3; 4 Milligram (mg) Baricitinib Phase 2; 4 mg Baricitinib Phase 3; Placebo Phase 2; Placebo Phase 3

SUMMARY:
This study is designed to select up to two doses of baricitinib (referred to as low dose and high dose) and assess their efficacy and safety for the treatment of severe or very severe alopecia areata. An additional subpopulation of 60 participants in the US will enroll in the open-label addenda.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years and ≤60 years for males (≤70 years of age for females) at the time of informed consent.
* Must self-identify as either Black or African American in race in the open label addenda.
* Have severe or very severe AA, as determined by all of the following:

  * Current AA episode of more than 6 months' duration and hair loss encompassing ≥50% of the scalp, as measured by -- SALT Alopecia Areata Investigator Global Assessment (AA-IGA) of 3 or 4) at screening and baseline.
  * No spontaneous improvement over the past 6 months.
  * Current episode of severe or very severe AA of less than 8 years.
  * Male or nonpregnant, nonbreastfeeding female participants.

Exclusion Criteria:

* Primarily "diffuse" type of AA.
* Are currently experiencing other forms of alopecia or any other concomitant conditions that would interfere with evaluations of the effect of study medication on AA.
* Previously treated with an oral Janus kinase (JAK) inhibitor and had an inadequate response (for example, absence of significant terminal hair growth after at least 12 weeks of treatment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Johnson Dermatology, Fort Smith, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Alliance Research Centers, Irvine, California
  - University of CA, Irvine, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Stanford Health Care, Redwood City, California
  - University of California Davis-Dermatology, Sacramento, California
  - University Clinical Trials, Inc., San Diego, California
  - Mosaic Dermatology, Santa Monica, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Medaphase Inc, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Forefront Research, Louisville, Kentucky
  - Callender Center for Clinical Research, LLC / Research, Glenn Dale, Maryland
  - ActivMed Practices and Research, Beverly, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clarkston Skin Research, Clarkston, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - ActivMed Practices and Research, Portsmouth, New Hampshire
  - University of Rochester School of Medicine, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OH State Univ College of Med, Gahanna, Ohio
  - NW Dermatology & Research Center, LLC, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - Penn State Univ. Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bellaire Dermatology, Bellaire, Texas
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Dermatology Associates, Seattle, Washington
- Japan (4):
  - Kurume University Hospital, Kurume, Fukuoka
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Tokyo Medical Univ. Hospital, Shinjuku-ku, Tokyo
  - Osaka City University Hospital, Osaka
- Mexico (8):
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Consultorio Privado de la Dra. Villanueva, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, N.L.
  - CRI Centro Regiomontano de Investigacion S.C., Monterrey, Nuevo León
  - B&B Investigaciones Medicas, SC, Mazatlán, Sinaloa
  - Derma Norte del Bajío, S.C., Aguascalientes
  - RM Pharma Specialists S.A. de C.V., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
- Puerto Rico (2):
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group, PSC- Hato Rey, San Juan, PR
- South Korea (11):
  - Seoul National University Bundang Hospital, Seongnam, Geonggi-do
  - Inha University Hospital, Jung-gu, Incheon
  - Chonbuk National University Hospital, Jeonju, Jeon Ra Buk-Do, Korea
  - Pusan National University Hospital, Busan, Korea
  - Kyung Pook National University Hospital, Daegu, Korea
  - Chungnam National University Hospital, Daejeon, Korea
  - Seoul National University Hospital, Seoul
  - Eunpyeong St. Mary's Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Chungang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] King B, Mostaghimi A, Shimomura Y, Piraccini BM, Blume-Peytavi U, Sontag A, Dutronc Y, Denning K, Kolodsick J, Lu X, Srivastava A, Sinclair R. Safety of Baricitinib in Adults with Severe Alopecia Areata from Two Phase III Trials Over a Median of 2.3 Years and Up to 4 Years of Treatment. Am J Clin Dermatol. 2025 Jul;26(4):611-622. doi: 10.1007/s40257-025-00932-0. Epub 2025 Apr 11. PMID 40214720
- [Derived] King B, Ko J, Kwon O, Vano-Galvan S, Piraccini BM, Dutronc Y, Yu G, Liu C, Somani N, Ball S, Mesinkovska NA. Baricitinib Withdrawal and Retreatment in Patients With Severe Alopecia Areata: The BRAVE-AA1 Randomized Clinical Trial. JAMA Dermatol. 2024 Oct 1;160(10):1075-1081. doi: 10.1001/jamadermatol.2024.2734. PMID 39141364
- [Derived] Craiglow B, Lee YW, Vano-Galvan S, Egeberg A, Dutronc Y, Durand F, Pierce E, Yu G, Chen YF, Mostaghimi A. Improvement in Measures of Quality of Life and Symptoms of Anxiety and Depression in Patients with Severe Alopecia Areata Achieving Sustained Scalp Hair Regrowth with Baricitinib. Dermatol Ther (Heidelb). 2024 Jul;14(7):1959-1968. doi: 10.1007/s13555-024-01208-x. Epub 2024 Jun 21. PMID 38904749
- [Derived] Senna MM, Kwon O, Piraccini BM, Sinclair R, Ball S, Ding Y, Chen YF, Dutronc Y, King B. Clinical Benefits of Baricitinib Therapy According to Scalp Hair Regrowth in Patients with Severe Alopecia Areata. Dermatol Ther (Heidelb). 2023 Dec;13(12):3209-3220. doi: 10.1007/s13555-023-01063-2. Epub 2023 Nov 22. PMID 37991697
- [Derived] Ko JM, Mayo TT, Bergfeld WF, Dutronc Y, Yu G, Ball SG, Somani N, Craiglow BG. Clinical Outcomes for Uptitration of Baricitinib Therapy in Patients With Severe Alopecia Areata: A Pooled Analysis of the BRAVE-AA1 and BRAVE-AA2 Trials. JAMA Dermatol. 2023 Sep 1;159(9):970-976. doi: 10.1001/jamadermatol.2023.2581. PMID 37556146
- [Derived] Piraccini BM, Ohyama M, Craiglow B, Bewley A, Ding Y, Chen YF, Dutronc Y, Pierce E, Durand F, Mostaghimi A. Scalp hair regrowth is associated with improvements in health-related quality of life and psychological symptoms in patients with severe alopecia areata: results from two randomized controlled trials. J Dermatolog Treat. 2023 Dec;34(1):2227299. doi: 10.1080/09546634.2023.2227299. PMID 37381691
- [Derived] Kwon O, Senna MM, Sinclair R, Ito T, Dutronc Y, Lin CY, Yu G, Chiasserini C, McCollam J, Wu WS, King B. Efficacy and Safety of Baricitinib in Patients with Severe Alopecia Areata over 52 Weeks of Continuous Therapy in Two Phase III Trials (BRAVE-AA1 and BRAVE-AA2). Am J Clin Dermatol. 2023 May;24(3):443-451. doi: 10.1007/s40257-023-00764-w. Epub 2023 Mar 1. PMID 36855020
- [Derived] King B, Mostaghimi A, Shimomura Y, Zlotogorski A, Choi GS, Blume-Peytavi U, Passeron T, Holzwarth K, Dutronc Y, McCollam J, Yang FE, Stanley S, Wu WS, Sinclair R. Integrated safety analysis of baricitinib in adults with severe alopecia areata from two randomized clinical trials. Br J Dermatol. 2023 Feb 10;188(2):218-227. doi: 10.1093/bjd/ljac059. PMID 36763878
- [Derived] King B, Ohyama M, Kwon O, Zlotogorski A, Ko J, Mesinkovska NA, Hordinsky M, Dutronc Y, Wu WS, McCollam J, Chiasserini C, Yu G, Stanley S, Holzwarth K, DeLozier AM, Sinclair R; BRAVE-AA Investigators. Two Phase 3 Trials of Baricitinib for Alopecia Areata. N Engl J Med. 2022 May 5;386(18):1687-1699. doi: 10.1056/NEJMoa2110343. Epub 2022 Mar 26. PMID 35334197
- See also: A Study of Baricitinib (LY3009104) in Participants With Severe or Very Severe Alopecia Areata (Hair Loss) — https://trials.lilly.com/ext/trial?id=I4V-MC-JAHO

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was divided into 2 stages separated by a decision point for Phase 3 dose selection, after all patients from the Phase 2 portion of the study had completed 12 weeks of treatment or had discontinued early. Approximately 100 patients were planned to be enrolled in the Phase 2 portion of the study. The remaining approximately 625 patients were planned to be enrolled into the Phase 3 portion.
Pre-assignment Details: After Decision Point participants randomized during Stage 1 to 1 mg Baricitinib were transitioned to the 4 mg Baricitinib.
  Results up to Week 36 (primary outcome) are reported here; data beyond Week 36, including open-label addenda, will be reported with the final results.
Groups:
- Placebo Phase 2: Participants received three placebo tablets administered orally every day (QD).
- 1 Milligram (mg) Baricitinib Phase 2: Participants received one 1 mg Baricitinib tablet administered orally QD, and two placebo tablets administered orally QD to maintain the blind.
- 4 mg Baricitinib Phase 2: Participants received one 4 mg Baricitinib tablet administered orally, QD and two placebo tablets QD administered orally to maintain the blind.
Period: Overall Study
Arm/Group | Placebo Phase 2 | 1 Milligram (mg) Baricitinib Phase 2 | 2 mg Baricitinib Phase 2 | 4 mg Baricitinib Phase 2 | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Started | 28 | 28 | 27 | 27 | 189 | 184 | 281
Received at Least One Dose of Study Drug | 28 | 28 | 27 | 27 | 189 | 183 | 280
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 28 | 28 | 27 | 27 | 189 | 184 | 281
Not completed — Ongoing | 26 | 25 | 25 | 26 | 140 | 142 | 220
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 3 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 8 | 2 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 5 | 10 | 10
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Screen Fail | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 1 | 17 | 12 | 15
Not completed — Other | 0 | 0 | 0 | 0 | 17 | 14 | 21

BASELINE CHARACTERISTICS:
Population: The first approximately 100 randomized and treated participants in Phase 2 portion who completed Visit 8 (Week 36) assessment or discontinued early. All participants enrolled in Phase 3 portion, and who are randomized to baricitinib 4-mg, baricitinib 2-mg, and placebo treatment arms in both Stages 1 and 2.
Groups:
- 4 mg Baricitinib Phase 2: Participants received one 4 mg Baricitinib tablet administered orally, QD and two placebo tablet administered orally QD to maintain the blind.
- 4 mg Baricitinib Phase 3: Participants received one 4 mg Baricitinib tablet administered orally, QD and one placebo tablet QD administered orally to maintain the blind.
- Total: Total of all reporting groups
Arm/Group | Placebo Phase 2 | 1 mg Baricitinib Phase 2 | 2 mg Baricitinib Phase 2 | 4 mg Baricitinib Phase 2 | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3 | Total
Number analyzed (Participants) | 28 | 28 | 27 | 27 | 189 | 184 | 281 | 764
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed includes only participants with observed (non-missing) data for each specific baseline characteristic. In the 4 mg Baricitinib Phase 3 arm, age data for one participant was not collected and therefore couldn't be reported.
  years
    number analyzed (Participants) | 28 | 28 | 27 | 27 | 189 | 184 | 280 | 763
    (all) | 40.5 (14.23) | 38.6 (11.26) | 42.5 (13.75) | 42.4 (14.91) | 37.4 (12.91) | 38.0 (12.78) | 36.3 (13.27) | 41.0 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 23 | 25 | 109 | 109 | 165 | 465
  Male | 12 | 10 | 4 | 2 | 80 | 75 | 116 | 299
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 8 | 5 | 8 | 22
  Asian | 3 | 4 | 3 | 4 | 78 | 76 | 114 | 282
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Black or African American | 4 | 2 | 3 | 3 | 17 | 7 | 28 | 64
  White | 21 | 22 | 20 | 19 | 83 | 93 | 123 | 381
  More than one race | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 0 | 0 | 0 | 70 | 70 | 107 | 247
  United States | 25 | 25 | 24 | 24 | 103 | 102 | 153 | 456
  Japan | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 12
  Mexico | 0 | 0 | 0 | 0 | 16 | 12 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 20 - Phase 3
Description: The SALT uses a visual aid showing the division of the scalp hair into 4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score, as developed by the National Alopecia Areata Foundation Working Committee. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process. The SALT score will range from 0% to 100%, with lower score indicating better health outcomes.
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo Phase 3: Participants received two placebo tablets administered orally every day (QD).
- 4 mg Baricitinib Phase 3: Participants received one 4 mg Baricitinib tablet administered orally, every day QD, and one placebo tablet administered orally QD to maintain the blind.
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 189 | 184 | 281
percentage of participants | 5.3 [2.9 to 9.5] | 21.7 [16.4 to 28.2] | 35.2 [29.9 to 41.0]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.75, 95% CI 2-sided [2.75 to 12.02]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.80, 95% CI 2-sided [5.89 to 23.62]

2. Secondary Outcome: Percentage of Participants With Patient Reported Outcome (PRO) for Scalp Hair Assessment Score of 0 or 1 With a ≥ 2 Point Improvement From Baseline Among Participants With a Score of ≥ 3 at Baseline - Phase 3
Description: PRO is an assessment of the participant's current extent of scalp involvement. It is comprised of 5 category response options: 0= No missing hair (0% of my scalp is missing hair; I have a full head of hair); 1 = A limited area (1% to 20% of my scalp is missing hair); 2 = A moderate area (21% to 49% of my scalp is missing hair); 3 = A large area (50% to 94% of my scalp is missing hair); and 4 = Nearly all or all (95% to 100% of my scalp is missing hair).
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2 with baseline PRO for scalp hair assessment of ≥ 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 181 | 175 | 275
percentage of participants | 5.0 [2.6 to 9.2] | 16.0 [11.3 to 22.2] | 33.1 [27.8 to 38.9]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.81 to 8.51]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.26, 95% CI 2-sided [5.05 to 20.87]

3. Secondary Outcome: Percentage of Participants Achieving PRO Measure for EB 0 or 1 With ≥ 2-point Improvement From Baseline (Among Participants With PRO Measure for EB ≥ 2 at Baseline) - Phase 3
Description: PRO is an assessment of the participant's current appearance of eyebrows. It is comprised of 4 category response options: 0 = I have full EB on each eye; 1= I have a minimal gap(s) or a minimal amount of thinning in at least 1 of my EB; 2 = I have a large gap(s) or a large amount of thinning in at least 1 of my EB; and 3 = I have no or barely any EB hairs.
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2 with baseline PRO measure for EB ≥ 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 130 | 141 | 184
percentage of participants | 3.1 [1.2 to 7.6] | 16.3 [11.1 to 23.3] | 32.1 [25.7 to 39.1]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 5.58, 95% CI 2-sided [1.97 to 15.83]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.34, 95% CI 2-sided [5.30 to 38.83]

4. Secondary Outcome: Percentage of Participants Achieving PRO Measure for EL 0 or 1 With ≥ 2-point Improvement From Baseline (Among Participants With PRO Measure EL ≥2 at Baseline) - Phase 3
Description: PRO assessment of the participant's current appearance of EL. It is comprised of 4 category response options: 0 = I have full EL on each eyelid; 1 = I have a minimal gap or minimal gaps along the eyelids; 2 = I have a large gap or large gaps along the eyelids; and 3 = I have no or barely any EL hair.
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2 with baseline PRO measure for EL ≥ 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 100 | 112 | 161
percentage of participants | 2.0 [0.6 to 7.0] | 19.6 [13.3 to 28.0] | 29.8 [23.3 to 37.3]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.34, 95% CI 2-sided [2.72 to 39.30]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 18.47, 95% CI 2-sided [5.04 to 67.68]

5. Secondary Outcome: Percentage of Participants Achieving Clinician Reported Outcome (ClinRO) Measure for EyeBrow (EB) Hair Loss 0 or 1 With ≥ 2-point Improvement From Baseline (Among Participants With ClinRO Measure for EB Hair Loss ≥ 2 at Baseline) - Phase 3
Description: ClinRO is a clinician reported assessment which measures a participant's EB hair loss. It is comprised of 4 category response options: 0 = EB have full coverage and no areas of hair loss; 1 = There are minimal gaps in EB hair and distribution is even; 2 = There are significant gaps in EB hair or distribution is not even; 3 = No notable EB.
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2 with baseline ClinRO measure for EB Hair Loss ≥ 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 4 mg Baricitinib Phase: Participants received one 4 mg Baricitinib tablet administered orally QD, and one placebo tablet administered orally QD to maintain the blind.
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase
Number analyzed (Participants) | 124 | 136 | 188
percentage of participants | 3.2 [1.3 to 8.0] | 19.1 [13.4 to 26.5] | 31.4 [25.2 to 38.3]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.60, 95% CI 2-sided [2.34 to 18.62]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.58, 95% CI 2-sided [5.01 to 36.81]

6. Secondary Outcome: Percentage of Participants Achieving ClinRO Measure for Eye Lash (EL) Hair Loss 0 or 1 With ≥ 2-point Improvement From Baseline (Among Participants With ClinRO Measure for EL Hair Loss ≥ 2 at Baseline) - Phase 3
Description: ClinRO measure for EL hair loss is comprised of 4 category response options: 0 = The EL form a continuous line along the eyelids on both eyes; 1 = There are minimal gaps and the EL are evenly spaced along the eyelids on both eyes; 2 = There are significant gaps along the eyelids or the EL are not evenly spaced along the eyelids; 3 = No notable EL.
Time Frame: Week 36
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2 with baseline ClinRO measure for EL hair loss ≥ 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 96 | 111 | 167
percentage of participants | 3.1 [1.1 to 8.8] | 13.5 [8.4 to 21.1] | 33.5 [26.8 to 41.0]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 4.63, 95% CI 2-sided [1.41 to 15.27]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.42, 95% CI 2-sided [4.73 to 43.93]

7. Secondary Outcome: Percent Change From Baseline in SALT Score - Phase 3
Description: The SALT uses a visual aid showing the division of the scalp hair into 4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score, as developed by the National Alopecia Areata Foundation Working Committee. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process. The SALT score will range from 0% to 100, with lower score indicating worse health outcomes. Least Squares Mean (LSM) was calculated using analysis of covariance (ANCOVA) with geographic region duration of current episode at baseline (< 4 years versus ≥4 years), treatment group, and baseline value in the model.
Time Frame: Baseline, Week 36
Population: All randomized participants in Phase 3 portion, Stages 1 and 2 with a nonmissing baseline and least one postbaseline measures. A modified last observation carried forward (mLOCF) imputation technique was used to replace missing data with the most recent non-missing post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 185 | 180 | 278
percent change | -8.13 (3.100) | -31.23 (3.157) | -45.79 (2.663)
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -23.10, 95% CI 2-sided [-30.57 to -15.63], Standard Error of Mean 3.806
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -37.65, 95% CI 2-sided [-44.24 to -30.89], Standard Error of Mean 3.447

8. Secondary Outcome: Percentage of Participants Achieving 50% Improvement of SALT (SALT50) - Phase 3
Description: SALT uses a visual aid showing the division of the scalp hair into 4 areas with the top of the head constituting 40% of total surface, the posterior/back of head 24%, right side and left side of head 18% each. The percentage of hair loss in each area is determined and is multiplied by the percentage of scalp covered by that area. The total sum of the 4 products of each area will give the SALT score, as developed by the National Alopecia Areata Foundation Working Committee. Only terminal hair is included in the SALT; vellus hair or any fine downy hair is not taken into account in the SALT scoring process . The SALT score will range from 0% to 100%. with lower score indicating better health outcomes.
Time Frame: Week 12
Population: All randomized participants in Phase 3 portion, in both Stages 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo Phase 3: Participants received two placebo tablets administered orally every day QD.
- 4 mg Baricitinib Phase 3: Participants received one 4 mg Baricitinib tablet administered orally every day QD, and one placebo tablet administered orally QD to maintain the blind.
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 189 | 184 | 281
percentage of participants | 4.8 [2.5 to 8.8] | 9.8 [6.3 to 14.9] | 21.7 [17.3 to 26.9]
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p = 0.047, Regression, Logistic; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.01 to 5.29]
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.03, 95% CI 2-sided [2.91 to 12.51]

9. Secondary Outcome: Time for Participants to Achieve SALT ≤ 20
Description: Time for participants to achieve SALT ≤ 20
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2026-01

10. Secondary Outcome: Mean Change From Baseline in Hospital Anxiety Depression Scale (HADS) Anxiety Score - Phase 3
Description: The Hospital Anxiety Depression Scale (HADS) is a 14 item self-assessment scale that determines the levels of anxiety and depression that a patient is experiencing over the past week. The HADS utilizes a 4-point Likert scale (e.g., 0 to 3) for each question and is intended for ages 12 to 65 years. Scores for each domain (anxiety and depression) can range from 0 to 21, with higher scores indicating greater anxiety or depression.
  LS mean was calculated using an ANCOVA model which includes geographic region, duration of current episode at baseline (<4 years vs. ≥4 years), treatment group and baseline score as fixed factors.
Time Frame: Baseline, Week 36
Population: All randomized participants in Phase 3 portion, Stages 1 and 2 with a nonmissing baseline and at least one postbaseline measure. The method used to handle missing data will be mLOCF which used the most recent nonmissing postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 177 | 174 | 272
score on a scale | -0.40 (0.234) | -1.22 (0.236) | -0.93 (0.199)
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.38 to -0.25], Standard Error of Mean 0.288
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p = 0.040, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.05 to -0.02], Standard Error of Mean 0.261

11. Secondary Outcome: Mean Change From Baseline in HADS Depression Score - Phase 3
Description: The HADS is a 14 item self-assessment scale that determines the levels of anxiety and depression that a patient is experiencing over the past week. The HADS utilizes a 4-point Likert scale (e.g., 0 to 3) for each question and is intended for ages 12 to 65 years. Scores for each domain (anxiety and depression) can range from 0 to 21, with higher scores indicating greater anxiety or depression.
  LS mean was calculated using an ANCOVA model which includes geographic region, duration of current episode at baseline (<4 years vs. ≥4 years), treatment group and baseline score as fixed factors.
  .
Time Frame: Baseline, Week 36
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
Number analyzed (Participants) | 177 | 174 | 272
score on a scale | 0.04 (0.210) | -0.38 (0.213) | -0.28 (0.179)
Statistical Analysis 1: Comparison: Placebo Phase 3 vs 2 mg Baricitinib Phase 3; Test type: Superiority; p = 0.107, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.93 to 0.09], Standard Error of Mean 0.259
Statistical Analysis 2: Comparison: Placebo Phase 3 vs 4 mg Baricitinib Phase 3; Test type: Superiority; p = 0.174, ANCOVA; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.78 to 0.14], Standard Error of Mean 0.234

ADVERSE EVENTS:
Time Frame: Baseline up to Week 36
Description: * All randomized participants who received at least one dose of the study drug and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first post-baseline visit.
  * Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo Phase 2: Participants received three placebo tablets administered QD.
- 1 mg Baricitinib Phase 2: Participants received one 1 mg Baricitinib tablet administered orally QD and two placebo tablets administered orally QD to maintain the blind.
- 2 mg Baricitinib Phase 2: Participants received one 2 mg Baricitinib tablet administered orally QD and two placebo tablets administered orally QD to maintain the blind.
- 4 mg Baricitinib Phase 2: Participants received one 4 mg Baricitinib tablet administered orally QD, and two placebo tablets QD administered orally to maintain the blind.
Arm/Group | Placebo Phase 2 | 1 mg Baricitinib Phase 2 | 2 mg Baricitinib Phase 2 | 4 mg Baricitinib Phase 2 | Placebo Phase 3 | 2 mg Baricitinib Phase 3 | 4 mg Baricitinib Phase 3
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/27 | 0/189 | 0/183 | 0/280
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/27 | 3/189 | 4/183 | 6/280
Other Adverse Events (participants affected / at risk) | 11/28 | 8/28 | 16/27 | 14/27 | 26/189 | 28/183 | 62/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Phase 2 (N=28) | 1 mg Baricitinib Phase 2 (N=28) | 2 mg Baricitinib Phase 2 (N=27) | 4 mg Baricitinib Phase 2 (N=27) | Placebo Phase 3 (N=189) | 2 mg Baricitinib Phase 3 (N=183) | 4 mg Baricitinib Phase 3 (N=280)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/16 (0) | 0/18 (0) | 0/23 (0) | 0/25 (0) | 0/109 (0) | 0/108 (0) | 1/164 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Phase 2 (N=28) | 1 mg Baricitinib Phase 2 (N=28) | 2 mg Baricitinib Phase 2 (N=27) | 4 mg Baricitinib Phase 2 (N=27) | Placebo Phase 3 (N=189) | 2 mg Baricitinib Phase 3 (N=183) | 4 mg Baricitinib Phase 3 (N=280)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 12 (12) | 12 (14) | 21 (28)
Onychomycosis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (8) | 1 (1) | 3 (3) | 5 (5) | 10 (13) | 9 (12) | 21 (29)
Vulvovaginal candidiasis (Infections and infestations) | 0/16 (0) | 1/18 (1) | 0/23 (0) | 0/25 (0) | 0/109 (0) | 0/108 (0) | 0/164 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/16 (1) | 0/18 (0) | 0/23 (0) | 0/25 (0) | 0/109 (0) | 0/108 (0) | 0/164 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1/16 (1) | 0/18 (0) | 0/23 (0) | 0/25 (0) | 0/109 (0) | 0/108 (0) | 0/164 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/16 (0) | 1/18 (1) | 0/23 (0) | 0/25 (0) | 0/109 (0) | 0/108 (0) | 0/164 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 10 (10) | 16 (18)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03570749/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03570749/SAP_003.pdf